CLINICAL TRIAL: NCT07347470
Title: Dancing Eyes: The Effect of Rhythmic Auditory Stimulation on VOR Gain Adaptation Among Healthy Adults - A Randomized Clinical Trial
Brief Title: The Effect of Rhythmic Auditory Stimulation on VOR Gain Adaptation Among Healthy Adults - A Randomized Clinical Trial "VOR - Vestibulo-ocular Reflex"
Acronym: VOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SMC-0074-23
Record Dates: First submitted 2025-12-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Vestibular adaptation
MeSH Terms: interventions — SIR1 protein, S cerevisiae

STUDY DESIGN:
Intervention Model Description: Participants will undergo vestibular adaptation training in 3 different conditions at least 48 hours apart - Silence, Metronome, and Music. the order will be randomly allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Silence (Active Comparator): Complete 15 minutes of vestibular adaptation training in silent condition
  Interventions: Other: Silence
- Metronome (Experimental): 15 minutes of vestibular adaptation training with metronome beat played in the background
  Interventions: Other: Rhythmic auditory stimulation
- Music (Experimental): 15 minutes of vestibular adaptation training with music played in the background
  Interventions: Other: Rhythmic auditory stimulation

INTERVENTIONS:
Other: Rhythmic auditory stimulation — the same 15 minutes of vestibular adaptation training will be completed by all participants in 3 different conditions: silence, metronome, and music. participants will be instructed to synchronize their head impulses to the beat in the auditory conditions.
  Arms: Metronome; Music
Other: Silence — 15 minutes of vestibular adaptation training without any background noise.
  Arms: Silence

SUMMARY:
The goal of this study is to learn whether adding rhythmic sound (a metronome beat or music) to eye-head exercises can improve the reflex that keeps vision clear during head movement. This reflex, called the vestibulo-ocular reflex (VOR), helps maintain visual stability during activities such as walking, turning, or bending. This type of training may help people with dizziness or balance problems, but this study focuses on healthy adults.

The main questions addressed are:

Does performing VOR exercises with a steady metronome beat improve the VOR more than performing the same exercises in silence?

Does performing the exercises while listening to self-selected rhythmic music also improve the VOR, and is the effect better or worse than a metronome?

Do the different sound conditions change how difficult the training feels or how dizzy participants feel?

Three conditions will be compared:

Silence: standard VOR training with no sound Metronome: training timed to a simple, steady beat Music: training performed while listening to self-selected music with a clear beat

The study will assess whether adding rhythmic sound leads to greater improvement in VOR gain and whether one type of sound is more effective than another.

Participants are healthy adults. Participants will:

Attend the laboratory for three separate visits, each with a different sound condition (silence, metronome, and music).

Visits will be at least 48 hours apart.

Wear specialized goggles that record eye and head movements (EyeSeeCam).

Perform brief eye-head tests before and after training, consisting of rapid head turns while maintaining fixation on a visual target.

Complete 15 minutes of Incremental VOR adaptation training during each visit, repeating rapid head turns while fixating on a laser projected target (StableEyes). In some sessions movements will be synchronized to a metronome or music.

Rate perceived training difficulty, ease of following the rhythm, and any dizziness or discomfort.

By comparing results across the three conditions within the same participants, the study will determine whether a simple, low-cost rhythmic cue can enhance the effects of standard VOR exercises without increasing discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Vestibular disorders. Neurologic conditions, Deafness, Blindness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in horizontal semicircular canal VOR gain for active and passive head impulses | Gains values- Baseline (pre-training) and immediately after each training session (post-training). Assessed during each of the three sessions. The sessions are separated by at least 48 hours and all three will be completed over approximately 2 - 4 weeks.
  The change in vestibulo-ocular reflex (VOR) gain for the horizontal semicircular canals, measured using video head impulse testing (vHIT), calculated as the difference between pre-training and post-training gain values for both active and passive head impulses under each auditory condition (Silence, Metronome, and Music).

SECONDARY OUTCOMES:
Self-reported training difficulty and adverse symptoms | Immediately after completion of each of the three training sessions. Sessions will be separated by at least 48 hours and all three will be completed over approximately 2-4 weeks.
  Participant-reported ratings of training difficulty and adverse symptoms (including dizziness and nausea), assessed using 1-10 visual analog scales completed after each training session under each of the three auditory conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel